CLINICAL TRIAL: NCT01595854
Title: Investigation of Pharmacodynamic Effects of Dabigatran and Ticagrelor (Part 1 and 2, Open, Non-randomised, 2 Parallel Groups) and Assessment of Ticagrelor Interaction Potential With Dabigatran (Part 3, Open, Randomised, Two-period Cross-over) in Healthy Male Subjects
Brief Title: Investigation of Pharmacodynamic Effects of Dabigatran and Ticagrelor and Assessment of Ticagrelor Interaction Potential With Dabigatran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.141; 2012-000874-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Ticagrelor

ARMS (4):
- Test 2 (part 3) (Experimental): low dose dabigatran + high dose ticagrelor
  Interventions: Drug: Ticagrelor; Drug: dabigatran etexilate
- Test 1 (part 1 + 2) (Active Comparator): high dose ticagrelor
  Interventions: Drug: Ticagrelor
- Reference 1 (part 1 + 2) (Experimental): medium dose dabigatran
  Interventions: Drug: dabigatran etexilate
- Reference 2 (part 3) (Experimental): low dose dabigatran
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — medium dose dabigatran
  Arms: Reference 1 (part 1 + 2)
Drug: Ticagrelor — high dose ticagrelor
  Arms: Test 1 (part 1 + 2)
Drug: Ticagrelor — high dose ticagrelor
  Arms: Test 2 (part 3)
Drug: dabigatran etexilate — low dose dabigatran
  Arms: Reference 2 (part 3)
Drug: dabigatran etexilate — medium dose dabigatran
  Arms: Test 2 (part 3)

SUMMARY:
Evaluation of potential ticagrelor effects on dabigatran exposure and evaluation of two new pharmacodynamic methods

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

   Exclusion criteria:
2. Any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.141.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran Etexilate 220 mg - Part 1: A single dose of dabigatran etexilate 220 mg (2 capsules of 110 mg), using a washed blood test.
- Ticagrelor 180 mg - Part 1: A single dose of ticagrelor coated tablets 180 mg (2 tablets of 90 mg), using a washed blood test.
- Dabigatran Etexilate 220 mg - Part 2: A single dose of dabigatran etexilate 220 mg (2 capsules of 110 mg), using a shed blood test.
- Ticagrelor 180 mg - Part 2: A single dose of ticagrelor coated tablets 180 mg (2 tablets of 90 mg), using a shed blood test
- Dabigatran Etexilate/Multiple Dose Ticagrelor Crossover-Part 3: A randomised, two-period, cross-over trial, the two treatments administered were
  * A single dose of dabigatran etexilate 75 mg
  * Ticagrelor coated tablets dosed for four days; 180 mg loading dose on day 1, 90 mg twice daily on day 2 and 3, 90 mg on day 4. Co-administered is a single dose of 75 mg Dabigatran etexilate on days 1 and 4.
  Between treatment periods there was a washout period of at least 4 days.
Period: Overall Study
Arm/Group | Dabigatran Etexilate 220 mg - Part 1 | Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 220 mg - Part 2 | Ticagrelor 180 mg - Part 2 | Dabigatran Etexilate/Multiple Dose Ticagrelor Crossover-Part 3
Started | 8 | 4 | 8 | 4 | 12
Completed | 8 | 4 | 8 | 4 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dabigatran Etexilate / Multiple Dose Ticagrelor - Part 3: A randomised two-period cross-over trial, the two treatments administered were
  * A single dose of dabigatran etexilate 75 mg
  * Ticagrelor coated tablets dosed for four days; 180 mg loading dose on day 1, 90 mg twice daily on day 2 and 3, 90 mg on day 4. Co-administered with a single dose of 75 mg Dabigatran etexilate on days 1 and 4.
  Between treatment periods there was a washout period of at least 4 days.
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate 220 mg - Part 1 | Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 220 mg - Part 2 | Ticagrelor 180 mg - Part 2 | Dabigatran Etexilate / Multiple Dose Ticagrelor - Part 3 | Total
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 12 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 30.6 (7.7) | 29.8 (11.4) | 33.6 (9.1) | 33.3 (6.3) | 30.2 (7.2) | 31.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 4 | 8 | 4 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Total Dabigatran (Dabi): Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma, over the time interval from 0 extrapolated to infinity, of dabigatran.
Time Frame: -1/-0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours
Population: Pharmacokinetic (PK) set defined as all subjects of Part 3 who received at least 1 dose of trial medication and provided at least 1 observation for at least 1 PK endpoint without important protocol violations relevant to the evaluation of bioavailability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Dabi 75 mg: A single dose of Dabigatran etexilate (Dabi) 75 mg.
- Dabi + Ticagrelor LD: A single dose of 75 mg Dabigatran coadministered with a loading dose (LD) of 180 mg ticagrelor coated tablets (T).
- Dabi + Ticagrelor MD: A single dose of 75 mg Dabigatran coadministered with a morning dose of multiple dose (MD) ticagrelor.
Arm/Group | Dabi 75 mg | Dabi + Ticagrelor LD | Dabi + Ticagrelor MD
Number analyzed (Participants) | 12 | 12 | 12
ng*h/mL | 281.05 (104) | 485.48 (40.5) | 410.46 (53.1)

2. Primary Outcome: Total Dabigatran: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of total dabigatran in plasma, per period.
Time Frame: -1/-0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dabi + Ticagrelor MD: A single dose of 75 mg Dabigatran coadministered with a morning dose of multiple dose (LD) ticagrelor.
Arm/Group | Dabi 75 mg | Dabi + Ticagrelor LD | Dabi + Ticagrelor MD
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 31.47 (130) | 61.30 (42.9) | 49.11 (64.8)

3. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: The number of participants with drug related adverse events
Time Frame: From screening until the end-of-study examination
Population: Treated set
Measure: Number; unit: participants
Groups:
- Dabigatran 220 mg - Part 1: A single dose of Dabigatran etexilate 220 mg (2 capsules of 110 mg), using a washed blood test.
- Dabigatran 220 mg - Part 2: A single dose of Dabigatran etexilate 220 mg (2 capsules of 110 mg), using a shed blood test.
- Dabigatran 75 mg - Part 3: A single dose of Dabigatran etexilate 75 mg
- Dabigatran + Ticagrelor - Part 3: Ticagrelor coated tablets dosed for four days; 180 mg loading dose on day 1, 90 mg twice daily on day 2 and 3, 90 mg on day 4. Co-administered is a single dose of 75 mg Dabigatran etexilate on days 1 and 4.
Arm/Group | Dabigatran 220 mg - Part 1 | Ticagrelor 180 mg - Part 1 | Dabigatran 220 mg - Part 2 | Ticagrelor 180 mg - Part 2 | Dabigatran 75 mg - Part 3 | Dabigatran + Ticagrelor - Part 3
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 12 | 12
participants | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 to 10 days after last dosing
Groups:
- Dabi 75 mg - Part 3: A single dose of dabigatran etexilate (Dabi) 75 mg
- Multiple Dose Ticagrelor - Part 3: Ticagrelor coated tablets dosed for four days; 180 mg loading dose on day 1, 90 mg twice daily on day 2 and 3, 90 mg on day 4. Co-administered is a single dose of 75 mg Dabigatran etexilate on days 1 and 4.
Arm/Group | Dabigatran Etexilate 220 mg - Part 1 | Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 220 mg - Part 2 | Ticagrelor 180 mg - Part 2 | Dabi 75 mg - Part 3 | Multiple Dose Ticagrelor - Part 3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/8 | 0/4 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/8 | 0/4 | 0/8 | 0/4 | 2/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 220 mg - Part 1 (N=8) | Ticagrelor 180 mg - Part 1 (N=4) | Dabigatran Etexilate 220 mg - Part 2 (N=8) | Ticagrelor 180 mg - Part 2 (N=4) | Dabi 75 mg - Part 3 (N=12) | Multiple Dose Ticagrelor - Part 3 (N=12)
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.